CLINICAL TRIAL: NCT03956381
Title: A Study to Demonstrate the Accuracy of Femoral Neck Resection Compared to the Pre-operatively Selected OPS™ Plan in Total Hip Arthroplasty.
Brief Title: Accuracy of OPS™ Femoral Neck Resection Study
Status: Completed | Type: Observational
Sponsor: Corin (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP2018-03
Record Dates: First submitted 2019-05-08; First posted 2019-05-20 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Primary Total Hip Arthroplasty
Keywords: Femoral neck resection, offset, leg lenght, femoral anteversion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- THR with OPS system-TriFit TS/Trinity combination: Hip prosthesis combination: TriFit TS stem/ Trinity cup implanted by Surgeon 1 via a posterolateral approach according to their standard of practice.
  Interventions: Device: Primary Total Hip Replacement with Trinity cup and TriFit TS stem via posterolateral surgical approach.
- THR with OPS system-MetaFix/Trinity combination: Hip prosthesis combination: MetaFix stem/ Trinity cup implanted by Surgeon 2 via a direct anterior approach according to their standard of practice.
  Interventions: Device: Primary Total Hip Replacement with Trinity cup and MetaFix stem via direct anterior surgical approach

INTERVENTIONS:
Device: Primary Total Hip Replacement with Trinity cup and TriFit TS stem via posterolateral surgical approach. — The participant will undergo surgery using the hip prostheses and surgical approach used by their surgeon Investigator. A patient specific femoral guide, generated by the OPS™ plan preoperatively, will be used during the surgical step of femoral neck resection. These are not study specific procedures as the OPS™ system is already in use by the surgeon Investigator in their standard of practice.
  Groups: THR with OPS system-TriFit TS/Trinity combination
Device: Primary Total Hip Replacement with Trinity cup and MetaFix stem via direct anterior surgical approach — The participant will undergo surgery using the hip prostheses and surgical approach used by their surgeon Investigator. A patient specific femoral guide, generated by the OPS™ plan preoperatively, will be used during the surgical step of femoral neck resection. These are not study specific procedures as the OPS™ system is already in use by the surgeon Investigator in their standard of practice.
  Groups: THR with OPS system-MetaFix/Trinity combination

SUMMARY:
The primary objective of this study is to determine the accuracy of the Optimized Positioning System (OPS™) planning and delivery tools using different types of surgical approaches.

DETAILED DESCRIPTION:
Total Hip Replacement (THR) is the gold standard for treatment of severe arthritis of the hip as it relieves pain, restores function of the joint and improves quality of life for patients. The restoration of hip mechanics can be influenced by the selected femoral stem design and also by choices made by the surgeon during the surgical implantation. The combination of femoral neck resection level and angle are key factors, particularly in cementless hip arthroplasty, in determining post-operative leg length and femoral anteversion. Historically, an estimation of prosthesis sizing and positioning has been made via a process of manual or digital templating either pre or intraoperatively using images of the implants positioned over the standard AP and lateral view hip x-rays taken in advance of surgery with generic instruments used during the surgery to execute the femoral head resection at the planned level. This process has a number of limitations. The OPS™ system utilizes detailed pre-operative imaging including a CT scan to generate a plan for the femoral neck resection level and angulation based on the anatomy of the individual patient. Following validation of this plan by the operating clinician, a patient specific femoral guide instrument is generated to help facilitate the reliable delivery of the planned resection intraoperatively. The purpose of this study will be to evaluate the use of the patient-specific femoral instrument in the hands of two surgeons using different prosthesis combinations and surgical approaches. A total number of 40 participants will be enrolled. Participants in this study will return for a single post-operative visit at 6 weeks to have X-rays taken and to enable any post-operative study hip related complications to be recorded. Once this has been completed, participants will be routinely followed-up by their orthopaedic surgeon as required in accordance with standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who understand the conditions of the study and are willing to return to the clinical site at 6 weeks post-operatively.
2. Patients of either gender who are between 21-85 years inclusive.
3. Patients with a diagnosis of osteoarthritis, rheumatoid arthritis or osteonecrosis and are considered by the Investigator to be clinically and medically suitable to undergo a primary total hip replacement
4. Patients who meet the indications and none of the contraindications listed in the Instructions for Use (IFU) supplied by the manufacturer for the femoral stem and acetabular cup to be implanted.
5. Patients who meet the indications and none of the contraindications listed in the Instructions for Use (IFU) supplied by the manufacturer for OPS™ Femoral Plan and OPS™ Femoral Patient Specific Instruments.

Exclusion Criteria:

1. Patients who are unable to provide informed consent.
2. Patients who are unable to comply with all the required study procedures.
3. Patients whose insurance will not cover the cost of the pre-operative CT and functional x-ray imaging required for use of the OPS system.
4. Patients who are currently involved in any personal injury litigation, medical-legal or worker's compensations claims.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from the clinic registry at each of the investigational sites of those patients requiring a primary hip replacement. Those who meet the inclusion/exclusion criteria will be invited to enrol into the study.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of the final osteotomy level compared to the selected OPS™ plan preopertively. | 6 weeks post-op (+/- 2 weeks)
  Accuracy of the final osteotomy level compared to the selected OPS™ plan (+ or - 3mm). Two standard of care post-operative x-rays taken at 6 weeks will be used to evaluate the positioning of the total hip prosthesis from the resultant level of resection of the femoral neck. This parameter will be measured in mm.

SECONDARY OUTCOMES:
Comparison of the femoral stem size implanted compared to the selected OPS™ Plan preoperatively (± 1 size) | Immediate postoperative
  The femoral stem size used during the operation will be compared to the selected one by the OPS™ Plan. This parameter will be measured in units.
Comparison of the acetabular cup size implanted compared to the selected OPS™ Plan preoperatively. | Immediate postoperative
  The acetabular cup size used during the operation will be compared to the selected one by the OPS™ Plan. This parameter will be measured in mm.
Comparison of the femoral head size implanted compared to the selected OPS™ Plan preoperatively. | Immediate postoperative
  The femoral head size used during the operation will be compared to the selected one by the OPS™ Plan. This parameter will be measured in mm.
Measurement of any change in Leg length/ femoral head height compared to the preoperative OPS™ Plan (± 5mm). | 6 weeks post-op (+/- 2 weeks)
  The postoperative Leg length / femoral head height will be measured in mm and compared to the preoperative value.
Comparison of the acetabular cup orientation to the selected OPS™ Plan. | 6 weeks post-op (+/- 2 weeks)
  The planned versus achieved acetabular cup orientation will be measured using 2D/3D registration software, in degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Jennings, MD, Principal Investigator — Colorado Joint Replacement
Locations (1):
- Colorado Joint Replacement, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Optimized Positioning System (OPS™) — https://www.coringroup.com/uk/solutions/optimized-positioning-system-ops/